CLINICAL TRIAL: NCT03953183
Title: A Randomized, Double-blinded, 2-arm Parallel Groups, Single Center Study to Assess Product Use and Adaptation, Safety and Tolerability of P3P, a Novel Nicotine-containing Product, in Adult Healthy Cigarette Smokers Switching to One of Two P3P Variants for One Month
Brief Title: Product Use and Adaptation, Safety and Tolerability of P3P in Adult Healthy Smokers Switching to it
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: P3P-SE-02-RU
Record Dates: First submitted 2019-05-15; First posted 2019-05-16 (Actual); Results first posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-11

CONDITIONS: Pharmacokinetics
Keywords: Nicotine

STUDY DESIGN:
Intervention Model Description: A randomized, double-blinded, 2-arm parallel groups, single center study
Who Masked: Participant, Investigator
Masking Description: Neither the site staff nor the subject will be informed about the product variant the subjects have been randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P3P-1mg (Other): Subjects randomized to exclusive use of P3P-1mg
  Interventions: Other: P3P-1mg
- P3P-2mg (Other): Subjects randomized to exclusive use of P3P-2mg
  Interventions: Other: P3P-2mg

INTERVENTIONS:
Other: P3P-1mg — P3P-1mg (P3P product containing 1mg of nicotine.)
  Arms: P3P-1mg
Other: P3P-2mg — P3P-2mg (P3P product containing 2mg of nicotine.)
  Arms: P3P-2mg

SUMMARY:
The purpose of the study is to evaluate the product use and adaptation in adult, current cigarette smoking subjects between baseline and after one month of use of one of two P3P variants. The effect of P3P use behavior on nicotine pharmacokinetic (PK) profile, acceptability, as well as the safety and tolerability of P3P over a period of 1 month will be investigated.

DETAILED DESCRIPTION:
This is a study of daily use of up to 15 P3P products over one month, including 2 confinement periods (2 overnight stays at the beginning of the study and 1 overnight stay at the end of the exposure period). During the confinement visits, nicotine PK from P3P exposure will be assessed as well as pharmacodynamic effects related to craving, sensory parameters, product experience, and product acceptance.

Between the two confinement periods, subjects will return to the investigational site for weekly ambulatory visits during which P3P will be resupplied and selected safety and other study assessments will be performed.

From the start of the exposure period onwards, subjects will be instructed not to smoke or use other tobacco or nicotine containing products and to use P3P exclusively.

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed and dated the ICF and is able to understand the information provided in it.
* Subject has been a smoker for at least the last 3 years prior to the Screening Visit and has smoked 5 to 15 commercially available cigarettes per day for the last 3 months prior to Screening.
* Subject has a positive urinary cotinine test (cotinine ≥ 200 ng/mL).
* Subject does not plan to quit smoking within 2 months.
* Smoking, healthy subject as judged by the Investigator or designee based on available assessments from the Screening period.
* Ready to switch from smoking cigarettes to using P3P for the duration of the study.

Exclusion Criteria:

* As per the Investigator's judgment, the subject cannot participate in the study for any reason other than medical (e.g., psychological and/or social reason).
* Subject has a clinically relevant disease which requires medication or any other clinically significant medical condition, which as per the judgment of the Investigator would jeopardize the safety of the subject.
* Subject has asthma condition (post-bronchodilator FEV1/FVC < 0.75 and reversibility in FEV1 ≥ 12% and > 200 mL from pre- to post-bronchodilator values).
* Subject has (FEV1/FVC) < 0.7 and FEV1 < 80% predicted value at post-bronchodilator spirometry.
* Subject has a BMI < 18.5 kg/m2 or > 32.0 kg/m2.
* Subject has received medication within 14 days or within 5 half-lives of the drug prior to Admission (whichever is longer) which has an impact on CYP2A6 activity.
* Subject has a positive serology test for HIV 1/2, Hepatitis B, or Hepatitis C.
* Subject has a positive alcohol breath test and/or a history of alcohol disorder within the past 2 years.
* Subject has a positive urine drug test.
* Subject has participated in another clinical study within 3 months prior to the Screening Visit.
* Subject has been previously screened or enrolled in this study.
* For women only: subject is pregnant or is breastfeeding.
* For women of childbearing potential only: subject does not agree to use an acceptable method of effective contraception.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Haziza, PhD, Study Chair — Philip Morris Products SA; Vasilyuk V Bogdanovich, MD, Principal Investigator — LLC Scientific Research Center Eco-Safety
Locations (1):
- LLC Scientific Research Center Eco-Safety, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chrea C, Acquadro C, Afolalu EF, Spies E, Salzberger T, Abetz-Webb L, Cano S, Arnould B, Mainy N, Rose J, Weitkunat R. Developing fit-for-purpose self-report instruments for assessing consumer responses to tobacco and nicotine products: the ABOUT Toolbox initiative. F1000Res. 2018 Dec 2;7:1878. doi: 10.12688/f1000research.16810.1. eCollection 2018. PMID 30906527

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | P3P-1mg | P3P-2mg
Started | 30 | 30
Completed | 30 | 28
Not Completed | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | P3P-1mg | P3P-2mg | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.3 (4.82) | 30.0 (8.36) | 28.2 (7.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 17 | 17 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 30 | 30 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 174 (9.49) | 172 (12.5) | 173 (11.0)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.3 (3.69) | 24.0 (3.48) | 23.7 (3.58)

OUTCOME MEASURES:

1. Primary Outcome: Plasma Nicotine Concentration-time Profile
Description: To measure the plasma nicotine concentration-time profile following correction of baseline nicotine levels.
Time Frame: Derived from multiple blood sampling pre- and post-product use (over 4 hours post-product use), on day 1 and day 30.
Population: Some participants were excluded from analysis for protocol deviations. For participants in whom the elimination rate constant could not be calculated for any of the visits, background-corrected nicotine concentrations were considered as missing.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | P3P-1mg | P3P-2mg
Number analyzed (Participants) | 30 | 28
ng/ml
  4 mins after start of product use (Day 1) | 0.563 [0.384 to 0.824] | 0.563 [0.370 to 0.858]
  7 mins after start of product use (Day 1) | 0.928 [0.635 to 1.36] | 1.02 [0.688 to 1.51]
  10 mins after start of product use (Day 1) | 0.982 [0.699 to 1.38] | 1.39 [0.949 to 2.03]
  15 mins after start of product use (Day 1) | 1.18 [0.914 to 1.54] | 1.58 [1.14 to 2.20]
  30 mins after start of product use (Day 1) | 1.24 [0.969 to 1.60] | 1.59 [1.09 to 2.34]
  1 hr after start of product use (Day 1) | 1.07 [0.850 to 1.34] | 1.45 [1.04 to 2.02]
  2 hr after start of product use (Day 1) | 0.702 [0.546 to 0.904] | 1.08 [0.824 to 1.41]
  4 hr after start of product use (Day 1) | 0.353 [0.272 to 0.458] | 0.570 [0.416 to 0.781]
  4 mins after start of product use (Day 30) | 1.01 [0.784 to 1.31] | 0.990 [0.621 to 1.58]
  7 mins after start of product use (Day 30) | 1.28 [0.985 to 1.66] | 1.34 [0.866 to 2.08]
  10 mins after start of product use (Day 30) | 1.46 [1.19 to 1.78] | 1.62 [1.13 to 2.31]
  15 mins after start of product use (Day 30) | 1.45 [1.21 to 1.75] | 1.67 [1.13 to 2.46]
  30 mins after start of product use (Day 30) | 1.29 [1.01 to 1.65] | 1.76 [1.21 to 2.56]
  1 hr after start of product use (Day 30) | 1.16 [1.01 to 1.33] | 1.71 [1.29 to 2.26]
  2 hr after start of product use (Day 30) | 0.927 [0.726 to 1.18] | 1.16 [0.784 to 1.72]
  4 hr after start of product use (Day 30) | 0.530 [0.360 to 0.782] | 0.551 [0.361 to 0.840]

2. Primary Outcome: Maximum Nicotine Concentration [cCmax]
Description: To measure the maximum plasma nicotine concentration [cCmax] following correction of baseline nicotine levels.
Time Frame: Derived from multiple blood sampling pre- and post-product use (over 4 hours post-product use), on day 1 and day 30.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | P3P-1mg | P3P-2mg
Number analyzed (Participants) | 30 | 28
ng/mL
  Day 1 | 1.46 [1.12 to 1.89] | 2.11 [1.62 to 2.75]
  Day 30 | 2.05 [1.69 to 2.48] | 2.39 [1.73 to 3.32]

3. Primary Outcome: Time to the Maximum Nicotine Concentration [cTmax]
Description: To measure the time to maximum nicotine concentration [cTmax] following correction of baseline nicotine levels.
Time Frame: Derived from multiple blood sampling pre- and post-product use (over 4 hours post-product use), on day 1 and day 30.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | P3P-1mg | P3P-2mg
Number analyzed (Participants) | 30 | 28
minutes
  Day 1 | 30.0 [15.0 to 30.0] | 30.0 [15.0 to 30.0]
  Day 30 | 15.0 [10.0 to 30.0] | 30.0 [15.0 to 60.0]

4. Primary Outcome: Area Under the Concentration-time Curve From Start of Product Use (T0) to 4 Hours [cAUC(0-4h)]
Description: To measure the area under the plasma concentration-time curve [cAUC(0-4h)] following correction of baseline nicotine levels.
Time Frame: Derived from multiple blood sampling pre- and post-product use (over 4 hours post-product use), on day 1 and day 30.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hour/mL
Arm/Group | P3P-1mg | P3P-2mg
Number analyzed (Participants) | 30 | 28
ng*hour/mL
  Day 1 | 3.03 [2.34 to 3.92] | 4.74 [3.64 to 6.19]
  Day 30 | 3.96 [3.29 to 4.78] | 5.35 [3.85 to 7.43]

5. Secondary Outcome: Craving for a Cigarette
Description: Measured on a Visual Analogue Scale (VAS) of 0 (no craving) to 100 (strong craving). Over time results calculated as area under curve mm*hour.
Time Frame: Before, during and up to 4 hours post-product use on day 1 and day 30
Measure: Mean (95% Confidence Interval); unit: score on a scale (millimetres*hour)
Arm/Group | P3P-1mg | P3P-2mg
Number analyzed (Participants) | 30 | 28
score on a scale (millimetres*hour)
  Day 1 | 138 [111 to 166] | 111 [73.2 to 149]
  Day 30 | 130 [99.1 to 160] | 109 [68.6 to 149]

6. Secondary Outcome: Sensory Parameters
Description: Measured with a Sensory Questionnaire. Response to each question is assessed on a 7-point scale, ranging from 1 (not at all) to 7 (extremely).
Time Frame: Within 60 minutes after product use on day 1 and day 30.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | P3P-1mg | P3P-2mg
Number analyzed (Participants) | 30 | 29
score on a scale
  Puffs Evaluation/Liking (day 1) | 3.33 [2.82 to 3.85] | 3.50 [2.87 to 4.13]
  Puffs Harshness (day 1) | 4.60 [4.09 to 5.11] | 5.18 [4.74 to 5.61]
  Puffs Similar to Own Brand (day 1) | 2.33 [1.77 to 2.90] | 3.04 [2.24 to 3.83]
  Puffs Strength on Tongue (day 1) | 3.00 [2.47 to 3.53] | 3.57 [2.94 to 4.20]
  Puffs Strength in Nose (day 1) | 1.80 [1.40 to 2.20] | 2.07 [1.71 to 2.44]
  Puffs Strength in Back of Mouth/Throat (day 1) | 4.83 [4.30 to 5.36] | 5.07 [4.60 to 5.54]
  Puff Strength in Windpipe (day 1) | 4.50 [3.89 to 5.11] | 4.89 [4.44 to 5.34]
  Puff Strength in Chest (day 1) | 3.40 [2.78 to 4.02] | 3.86 [3.25 to 4.46]
  Puffs Evaluation/Liking (day 30) | 3.43 [2.97 to 3.90] | 3.46 [2.78 to 4.15]
  Puffs Harshness (day 30) | 4.20 [3.67 to 4.73] | 4.68 [4.15 to 5.21]
  Puffs Similar to Own Brand (day 30) | 2.93 [2.25 to 3.61] | 2.64 [2.04 to 3.24]
  Puffs Strength on Tongue (day 30) | 2.83 [2.26 to 3.41] | 3.36 [2.88 to 3.83]
  Puffs Strength in Nose (day 30) | 1.80 [1.43 to 2.17] | 1.93 [1.55 to 2.31]
  Puffs Strength in Back of Mouth/Throat (day 30) | 4.87 [4.31 to 5.43] | 4.86 [4.35 to 5.36]
  Puff Strength in Windpipe (day 30) | 4.20 [3.54 to 4.86] | 4.93 [4.45 to 5.41]
  Puff Strength in Chest (day 30) | 3.53 [2.89 to 4.17] | 4.07 [3.61 to 4.53]

7. Secondary Outcome: Product Experience
Description: Measured with ABOUT[TM]-Product Experience questionnaire. Response to each question is assessed on a 7-point scale, ranging from 1 (not at all) to 7 (extremely).
Time Frame: Within 60 minutes after product use on day 1 and day 30.
Measure: Mean (95% Confidence Interval); unit: score
Arm/Group | P3P-1mg | P3P-2mg
Number analyzed (Participants) | 30 | 29
score
  Aversion (day 1) | 1.25 [1.08 to 1.42] | 1.32 [1.12 to 1.53]
  Aversion (day 30) | 1.35 [1.10 to 1.60] | 1.45 [1.10 to 1.79]
  Craving reduction (day 1) | 4.23 [3.65 to 4.82] | 4.04 [3.38 to 4.69]
  Craving reduction (day 30) | 4.07 [3.47 to 4.66] | 4.14 [3.56 to 4.73]
  Psychological reward (day 1) | 3.00 [2.61 to 3.39] | 3.16 [2.66 to 3.65]
  Psychological reward (day 30) | 3.11 [2.72 to 3.49] | 2.93 [2.47 to 3.39]
  Enjoyment of respiratory tract sensations (day 1) | 2.13 [1.58 to 2.69] | 2.29 [1.65 to 2.92]
  Enjoyment of respiratory tract sensations (day 30) | 2.33 [1.81 to 2.86] | 2.29 [1.70 to 2.87]
  Product satisfaction (day 1) | 3.70 [3.26 to 4.14] | 3.62 [3.10 to 4.14]
  Product satisfaction (day 30) | 3.50 [3.06 to 3.94] | 3.42 [2.86 to 3.98]

8. Secondary Outcome: Product Dependence
Description: Measured with ABOUT[TM]-Dependence questionnaire. Response to each question is assessed on a 5-point scale, ranging from 1 (not at all/never) to 5 (extremely/all the time) or a 6-point scale ranging from 0 (more than 3 hours) to 5 (0-5 minutes).
Time Frame: Within 60 minutes after product use on day 1 and day 30.
Measure: Mean (95% Confidence Interval); unit: score
Arm/Group | P3P-1mg | P3P-2mg
Number analyzed (Participants) | 30 | 29
score
  Extent of use (day 1) | 57.9 [52.3 to 63.5] | 59.1 [52.9 to 65.2]
  Extent of use (day 30) | 52.8 [47.2 to 58.5] | 53.0 [47.4 to 58.6]
  Signs and symptoms (day 1) | 45.2 [42.1 to 48.4] | 49.5 [45.7 to 53.3]
  Signs and symptoms (day 30) | 38.3 [33.7 to 43.0] | 41.1 [37.4 to 44.8]
  Behavioral impact (day 1) | 32.3 [28.6 to 36.0] | 35.7 [30.2 to 41.2]
  Behavioral impact (day 30) | 23.5 [17.5 to 29.5] | 26.8 [20.9 to 32.6]

9. Secondary Outcome: Product Acceptance
Description: Measured with a Product Acceptance questionnaire. Response to each question is assessed on a 7-point scale, ranging from 1 (most negative) to 7 (most positive) or as multiple choice questions.
Time Frame: Within 60 minutes after product use on day 1 and day 30.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | P3P-1mg | P3P-2mg
Number analyzed (Participants) | 30 | 29
score on a scale
  Overall opinion about P3P (day 1) | 3.63 [3.10 to 4.17] | 3.46 [2.94 to 3.99]
  Overall opinion about P3P (day 30) | 3.80 [3.33 to 4.27] | 3.61 [2.88 to 4.33]
  Taste intensity (day 1) | 5.27 [4.65 to 5.88] | 5.36 [4.79 to 5.93]
  Taste intensity (day 30) | 5.03 [4.36 to 5.70] | 5.25 [4.52 to 5.98]
  Consistency of sensation (day 1) | 4.23 [3.81 to 4.66] | 3.93 [3.45 to 4.41]
  Consistency of sensation (day 30) | 3.93 [3.35 to 4.51] | 4.29 [3.78 to 4.79]
  Compared to pipe (day 1) | 4.00 [2.99 to 5.01] | 3.25 [2.10 to 4.40]
  Compared to pipe (day 30) | 3.77 [3.06 to 4.47] | 3.90 [2.71 to 5.09]
  Compared to hookah (day 1) | 3.28 [2.54 to 4.02] | 3.24 [2.36 to 4.11]
  Compared to hookah (day 30) | 3.40 [2.51 to 4.29] | 2.88 [1.84 to 3.92]
  Compared to heat-not-burn (day 1) | 3.27 [2.21 to 4.33] | 3.19 [1.92 to 4.45]
  Compared to heat-not-burn (day 30) | 3.06 [2.06 to 4.06] | 4.13 [2.99 to 5.28]
  Compared to e-cigarette (day 1) | 4.17 [3.21 to 5.12] | 3.76 [2.58 to 4.95]
  Compared to e-cigarette (day 30) | 3.71 [3.03 to 4.38] | 3.07 [2.07 to 4.07]
  Compared to snuff/chewing tobacco (day 1) | 5.00 [3.12 to 6.88] | 5.00 [2.09 to 7.91]
  Compared to snuff/chewing tobacco (day 30) | 3.56 [2.01 to 5.10] | 4.83 [2.59 to 7.08]
  Compared to NRT (day 1) | 6.40 [5.29 to 7.51] | 5.67 [3.21 to 8.12]
  Compared to NRT (day 30) | 4.86 [3.31 to 6.41] | 4.20 [1.51 to 6.89]

10. Secondary Outcome: Puffing Behavior of Subject
Description: To measure changes in subject puffing behavior. Evaluated by selection of one puffing behavior response out of three possible responses.
  * 1. Puffing and holding the aerosol in the mouth for a short time and then inhaling (i.e. like a cigarette)
  * 2. Puffing and immediately inhaling (without holding the aerosol in the mouth)
  * 3. Puffing and immediately exhaling, without inhalation
Time Frame: Evaluated by site staff on day 1 and day 30. Self-evaluated by subject on day 2, day 7, day 15, day 22, and day 29.
Measure: Count of Participants; unit: Participants
Arm/Group | P3P-1mg | P3P-2mg
Number analyzed (Participants) | 30 | 29
Participants
  Day 2: Inhalation Behavior #1 | 18 | 17
  Day 2: Behavior #2 | 12 | 11
  Day 2: Behavior #3 | 0 | 0
  Day 29: Behavior #1 | 20 | 21
  Day 29: Behavior #2 | 10 | 7
  Day 29: Behavior #3 | 0 | 0

11. Secondary Outcome: Overall Product Use
Description: To assess the number of any nicotine/tobacco products used overall on a daily basis.
Time Frame: Recorded daily by subject, in product use diary, from day 1 until day 30.
Measure: Mean (95% Confidence Interval); unit: products used per day
Arm/Group | P3P-1mg | P3P-2mg
Number analyzed (Participants) | 30 | 30
products used per day
  P3P | 6.54 [6.06 to 7.02] | 6.37 [5.54 to 7.21]
  Cigarettes | 2.64 [2.17 to 3.50] | 2.68 [1.84 to 3.52]
  Heat not burn and/or smokeless tobacco | 0.26 [-0.09 to 0.61] | 0.25 [-0.11 to 0.62]
  Other tobacco products | 0.02 [-0.02 to 0.06] | 0.01 [-0.01 to 0.03]
  Electronic cigarettes | 0.00 [-0.00 to 0.01] | 0.02 [-0.01 to 0.05]

12. Secondary Outcome: NEQ
Description: To measure percent changes from baseline in Nicotine equivalents (NEQ) concentrations, measured in spot urine and expressed as concentration adjusted for creatinine.
Time Frame: Measured at baseline, day 7, day 15, day 22, and day 29.
Population: Some participants were excluded from analysis for protocol deviations.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change from baseline
Arm/Group | P3P-1mg | P3P-2mg
Number analyzed (Participants) | 30 | 29
Percent change from baseline
  Day 7 | 20.3 [-11.5 to 52.1] | 30.1 [-16.7 to 76.8]
  Day 15 | 44.6 [-13.7 to 103] | 30.4 [0.0291 to 60.8]
  Day 22 | 41.7 [-16.0 to 99.3] | 18.8 [-1.89 to 39.5]
  Day 29 | 26.4 [-12.4 to 65.1] | 22.9 [-11.7 to 57.4]

13. Secondary Outcome: Total NNAL
Description: To measure percent changes from baseline in total 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL) concentrations, measured in spot urine and expressed as concentration adjusted for creatinine.
Time Frame: Measured at baseline, day 7, day 15, day 22, and day 29.
Population: Some participants were excluded from analysis for protocol deviations.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change from baseline
Arm/Group | P3P-1mg | P3P-2mg
Number analyzed (Participants) | 30 | 29
Percent change from baseline
  Day 7 | -7.07 [-46.9 to 32.8] | -17.1 [-36.3 to 2.05]
  Day 15 | -8.05 [-39.1 to 23.0] | -5.75 [-28.5 to 17.0]
  Day 22 | 14.3 [-27.9 to 56.4] | -14.4 [-33.6 to 4.75]
  Day 29 | -6.10 [-29.6 to 17.4] | -11.8 [-36.2 to 12.6]

14. Secondary Outcome: CEMA
Description: To measure percent changes from baseline in 2-cyanoethylmercapturic acid (CEMA) concentrations, measured in spot urine and expressed as concentration adjusted for creatinine (ng/mg creat).
Time Frame: Measured at baseline, day 7, day 15, day 22, and day 29.
Population: Some participants were excluded from analysis for protocol deviations.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change from baseline
Arm/Group | P3P-1mg | P3P-2mg
Number analyzed (Participants) | 30 | 29
Percent change from baseline
  Day 7 | -41.1 [-57.2 to -18.8] | -27.3 [-44.4 to -4.99]
  Day 15 | -38.5 [-55.7 to -14.5] | -26.0 [-46.3 to 2.08]
  Day 22 | -18.9 [-43.2 to 15.7] | -23.6 [-46.8 to 9.75]
  Day 29 | -28.3 [-52.9 to 9.07] | -30.8 [-50.2 to -3.87]

15. Secondary Outcome: CYP2A6 Activity
Description: To measure percent change from baseline in CYP2A6 enzymatic activity, on day 30, as measured by molar metabolic ratio of trans-3-hydroxy-cotinine/cotinine in plasma.
Time Frame: Measured before product use, on day 1 and day 30.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change from baseline
Arm/Group | P3P-1mg | P3P-2mg
Number analyzed (Participants) | 30 | 29
Percent change from baseline | 15.5 [-6.90 to 37.9] | 3.19 [-13.0 to 19.4]

16. Secondary Outcome: Amount of Powder Extracted From P3P Used for PK Assessment.
Description: Weight difference (mg) of P3P before and after use, to determine the amount of powder extracted from P3P.
Time Frame: Before and after product use, on day 1 and day 30.
Measure: Mean (95% Confidence Interval); unit: mg
Arm/Group | P3P-1mg | P3P-2mg
Number analyzed (Participants) | 30 | 28
mg
  Day 1 | 24.1 [20.7 to 27.4] | 22.4 [19.2 to 25.6]
  Day 30 | 28.9 [25.4 to 32.4] | 24.2 [19.8 to 28.6]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the signature of the ICF by each subject until the end of the safety follow-up period, for a total study duration of up to 45 days for each subject.
Arm/Group | P3P-1mg | P3P-2mg
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 7/30 | 5/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P3P-1mg (N=30) | P3P-2mg (N=30)
Blood Bilirubin Increased (Investigations) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specify that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belong to the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT03953183/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/83/NCT03953183/SAP_001.pdf